CLINICAL TRIAL: NCT02298010
Title: Pattern and Clinical Implication of Lymph Node Metastasis From Gastric Cancer Which Was Resected by Radical Surgery With Extended Lymphadenectomy
Brief Title: Lymph Node Metastasis in Extended Lymphadenectomy for Gastric Cancer From a CLASSIC Trial
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Saint Vincent's Hospital, Korea (Other); Gachon University Gil Medical Center (Other); Gangnam Severance Hospital (Other); Kyungpook National University Hospital (Other); Kyunghee University Medical Center (Other); Keimyung University Dongsan Medical Center (Other); Korea University Guro Hospital (Other); Korea University Anam Hospital (Other); Kosin University Gospel Hospital (Other); National Cancer Center, Korea (Other Government); Seoul Veterans Hospital (Other); Seoul National University Bundang Hospital (Other); Soonchunhyang University Hospital (Other); Severance Hospital (Other); Ajou University (Other); Yeungnam University Hospital (Other); Korea Cancer Center Hospital (Other); Ewha Womans University Mokdong Hospital (Other); Chonbuk National University Hospital (Other); Chonnam National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ML29471
Record Dates: First submitted 2014-11-19; First posted 2014-11-21 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2017-11

CONDITIONS: Stomach Neoplasms; Cancer of Lymph Node
MeSH Terms: conditions — Stomach Neoplasms | interventions — XELOX

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Adjuvant chemotherapy group: Research subjects who were enrolled in CLASSIC trial and underwent adjuvant chemotherapy.
  Interventions: Drug: Capecitabine, oxaliplatin
- Only surgery group: Research subjects who were enrolled in CLASSIC trial and did not undergo adjuvant chemotherapy

INTERVENTIONS:
Drug: Capecitabine, oxaliplatin
  Groups: Adjuvant chemotherapy group

SUMMARY:
The pattern of lymph node metastasis of the gastric cancer to each geographic lymph nose stations and the relation between each metastasis and survival are to be analyzed by retrospective review of medical records of who enrolled in the CLASSIC trial (NCT00411229) which have compared adjuvant chemotherapy and no adjuvant therapy after radical gastrectomy with extended lymphadenectomy.

ELIGIBILITY:
Criteria of previous CLASSIC trial:

Inclusion Criteria:

To be eligible for inclusion, each patient must fulfill each of the following criteria:

* Ambulatory males or females, aged ≥18 years.
* Karnofsky performance status of ≥70 %.
* Histologically confirmed gastric adenocarcinoma, staged pathologically, AJCC/UICC stage II (T2N1, T1N2, T3N0), IIIa (T3N1, T2N2, T4N0), and IIIb (T3N2). At least 15 examined lymph nodes are required to ensure the adequate TNM classification)
* Patients who underwent curative D2 lymphadenectomy resection for gastric cancer with no macroscopic or microscopic evidence for remaining tumor, who can be randomized to either study arm within 6 weeks after surgery.
* Give written informed consent prior to study specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.

Exclusion Criteria:

Patients who fulfill any of the following criteria will be excluded:

* Serious concomitant medical illnesses that would limit life expectancy to < 5 years.
* Pregnant or lactating women.
* Women of childbearing potential with either a positive or no pregnancy test at baseline. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-child bearing potential.
* Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study.
* Any evidence of metastatic disease (including presence of tumor cells in the ascites).
* Previous cytotoxic chemotherapy, radiotherapy or immunotherapy except corticosteroids, for the currently treated gastric cancer.
* History of another malignancy within the last five years except cured basal cell carcinoma of skin and cured carcinoma in-situ of uterine cervix.
* History of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the Investigator to be clinically significant precluding informed consent or interfering with compliance for oral drug intake.
* Clinically significant (i.e. active) cardiac disease e.g. symptomatic coronary artery disease, New York Heart Association (NYHA) grade II or greater congestive heart failure or serious cardiac arrhythmia requiring medication or myocardial infarction within the last 12 months.
* Lack of physical integrity of the upper gastrointestinal tract or those who have malabsorption syndrome likely to influence absorption of capecitabine, or inability to take oral medication.
* Known peripheral neuropathy ≥ CTCAEv3 grade 1. Absence of deep tendon reflexes (DTRs) as the sole neurologic abnormality does not render the patient ineligible.
* Organ allografts requiring immunosuppressive therapy.
* Serious uncontrolled intercurrent infections or other serious uncontrolled concomitant disease.-
* Moderate or severe renal impairment [creatinine clearance equal to or below 50 ml/min (calculated according to Cockroft and Gault)], or serum creatinine > 1.5 x upper limit of normal (ULN).
* Any of the following laboratory values:
* Absolute neutrophil count (ANC) < 1.5 x 10^9/L
* Platelet count < 100 x 10^9/L
* Total bilirubin > 1.5 x ULN
* ALAT, ASAT > 2.5 x ULN
* Alkaline phosphatase > 2.5 x ULN.
* Prior unanticipated severe reaction to fluoropyrimidine therapy (with or without documented DPD deficiency) or patients with Kknown dihydropyrimidine dehydrogenase (DPD) deficiency.
* Hypersensitivity to platinum compounds or any of the components of the study medications.
* Received any investigational drug or agent/procedure, i.e. participation in another trial, within 4 weeks before randomization.
* Blood transfusions or growth factors to aid hematologic recovery within 2 weeks prior to study treatment start.
* Requirement for concurrent use of the antiviral agent sorivudine (antiviral) or chemically related analogues, such as brivudine.
* Unwilling or unable to comply with the protocol for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study subjects who were enrolled in CLASSIC trial (NCT00411229) and whose medical records about the extent of the lymph node dissection and pathologic report are available.
Sampling Method: Non-Probability Sample
Enrollment: 899 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Topographic pattern of metastasis to regional lymph node stations | at the time of surgery

SECONDARY OUTCOMES:
survival according to the metastatic lymph node station | 3 and 5years
survival according to lymph node ratio | 3 and 5years
recurrence pattern | 3 and 5years